CLINICAL TRIAL: NCT05184712
Title: A Randomized, Double-blind, Multi-center, Phase III Study of AK112 Combined With Pemetrexed and Carboplatin Versus Placebo Combined With Pemetrexed and Carboplatin in Patients With Locally Advanced or Metastatic EGFR-mutant Non-squamous NSCLC Who Have Failed Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR-TKIs)
Brief Title: Phase 3 Clinical Study of AK112 for NSCLC Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-301; HARMONi-A (Other: Akeso)
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Non-Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — Injections; Pemetrexed; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ivonescimab (SMT112 or AK112) in combination with Pemetrexed and Carboplatin (Experimental): Subjects will receive Ivonescimab (SMT112 or AK112) Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles. Afterward, AK112 Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Interventions: Drug: Ivonescimab (SMT112 or AK112) Injection
- Placebo in combination with Pemetrexed and Carboplatin (Placebo Comparator): Subjects will receive Placebo Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles in treatment periods per the randomization schedule. Afterward, Placebo Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Interventions: Drug: Placebo Injection

INTERVENTIONS:
Drug: Ivonescimab (SMT112 or AK112) Injection — Subjects will receive Ivonescimab (SMT112 or AK112) Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles. Afterward, Ivonescimab (SMT112 or AK112) Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Other Names: Pemetrexed; Carboplatin
  Arms: Ivonescimab (SMT112 or AK112) in combination with Pemetrexed and Carboplatin
Drug: Placebo Injection — Subjects will receive Placebo Plus Pemetrexed and Carboplatin via intravenous infusion (IV) Q3W, up to 4 cycles in treatment periods per the randomization schedule. Afterward, Placebo Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.
  Other Names: Pemetrexed; Carboplatin
  Arms: Placebo in combination with Pemetrexed and Carboplatin

SUMMARY:
A Randomized, Double-blind, Multi-center, Phase III Clinical Study of AK112 or Placebo Combined With Pemetrexed and Carboplatin in Patients With EGFR-mutant Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Who Have Failed to Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) Treatment

DETAILED DESCRIPTION:
The trial will be performed as a randomized, Double-Blind, Multicenter trial to compare AK112 Plus Pemetrexed and Carboplatin to Placebo Plus Pemetrexed and Carboplatin in Patients with Locally Advanced or Metastatic Non-Squamous Non-Small Cell Lung Cancer (NSCLC) Harboring. Approximately 320 subjects will be randomized to the two treatment at the ratio of 1:1. Each enrolled subject will receive an intravenous infusion of the AK112/Placebo Plus Pemetrexed and Carboplatin （Q3W,up to 4 cycles）in treatment periods per the randomization schedule. Afterward, AK112/ Placebo Plus Pemetrexed will be used for maintenance treatment (administered on Day 1 of each cycle, Q3W) up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily sign a written informed consent form (ICF), which must be signed before the specified study procedures required for the study are performed.
2. Males or females aged ≥ 18 to ≤ 75 years at the time of signing informed consent.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1.
4. Life expectancy ≥3 months；
5. Locally advanced (stage IIIB/IIIC) or metastatic (stage IV) non-squamous NSCLC confirmed by histology or cytology, inoperable and unable to receive radiotherapy and chemotherapy;
6. The tumor histology, cytology or hematology confirmed the presence of EGFR activating mutations before enrollment
7. Have previously received EGFR-TKI treatment and the treatment has failed
8. Subjects have at least one measurable non-brain tumor lesion per RECIST v1.1
9. Major organ function prior to treatment meets the following criteria
10. Patients of childbearing potential must agree to use effective contraceptive measures

Exclusion Criteria:

1. Histological or cytological pathology confirmed the presence of small cell carcinoma components, or the main component is squamous cell carcinoma
2. There are reports confirming the existence of other driver gene mutations with known drug treatments
3. Subjects who received any prior treatments targeting the mechanism of tumor immunity
4. The subject has received systemic anti-tumor therapy other than EGFR-TKI
5. Currently enrolled in any other clinical study
6. Received EGFR-TKI treatment, palliative local treatment, non-specific immunomodulatory treatment within 2 weeks prior to the first dose; and Chinese herbal medicine or traditional Chinese medicinal products with anti-tumor indications within 1 weeks prior to the first dose.
7. Tumor surrounds important blood vessels or has obvious necrosis, cavitation, or invades surrounding important organs and blood vessels.
8. Symptomatic central nervous system metastases
9. Active malignancies within the past 3 years, with the exception of tumors in this study and cured local tumors
10. Active autoimmune disease requiring systemic treatment within 2 years prior to the start of study treatment
11. There is a history of major diseases 1 year prior to the first dose.
12. .Medical history of gastrointestinal perforation or gastrointestinal fistula within 6 months prior to the first dose
13. Received chest radiation therapy prior to the first dose
14. Presence of clinically symptomatic pleural effusion, pericardial effusion, or ascites requiring frequent drainage.
15. Active or previously documented inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival (PFS) assessed by IRC per RECIST v1.1 in the ITT population.

SECONDARY OUTCOMES:
OS | Up to 2 years
  Overall Survival (OS) in the ITT population
ORR | Up to 2 years
  Efficacy measures such as overall response rate (ORR), which is the proportion of subjects with CR or PR by IRRC based on RECIST v1.1
DCR | Up to 2 years
  Disease control rate (DCR), which is defined as the proportion of subjects with CR, PR, or SD, based on RECIST v1.1
DoR | Up to 2 years
  Duration of response (DoR), which is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
TTR | Up to 2 years
  TTR is defined as the time to response base on RECIST v1.1
PFS | Up to 2 years
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first assessed by investigator Per RECIST 1.1.
AE | From the subject signs the ICF to 30 days (AE) and 90 days (SAE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first,up to 2 years
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), and clinically significant abnormal laboratory results.
Observed concentrations of AK112 | through study completion, an average of 2 year
  The endpoints for assessment of PK of AK112 include serum concentrations of AK112 at different timepoints after AK112 administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK112 through 90 days after last dose of AK112,up to 2 years
  The immunogenicity of AK112 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] HARMONi-A Study Investigators; Fang W, Zhao Y, Luo Y, Yang R, Huang Y, He Z, Zhao H, Li M, Li K, Song Q, Du X, Sun Y, Li W, Xu F, Wang Z, Yang K, Fan Y, Liu B, Zhao H, Hu Y, Jia L, Xu S, Yi T, Lv D, Lan H, Li M, Liang W, Wang Y, Yang H, Jia Y, Chen Y, Lu J, Feng J, Liu C, Zhou M, Zhou J, Liu X, Zhou N, He M, Dong X, Chen H, Chen Y, Su H, Li X, Zhang Z, Yang L, Cheng Y, Chen L, Hou X, Zhang Y, Guo J, Wang Z, Lu H, Wu D, Feng W, Li W, Huang J, Wang Y, Song X, Peng J, Liu L, Guo Y, Li W, Lu D, Hu M, Wang ZM, Li B, Xia M, Zhang L. Ivonescimab Plus Chemotherapy in Non-Small Cell Lung Cancer With EGFR Variant: A Randomized Clinical Trial. JAMA. 2024 Aug 20;332(7):561-570. doi: 10.1001/jama.2024.10613. PMID 38820549